CLINICAL TRIAL: NCT01319851
Title: Alefacept and Allogeneic Hematopoietic Stem Cell Transplantation for Children With Non-Malignant Diseases Who Have Been Multiply Transfused: a Pilot Study
Brief Title: Alefacept and Allogeneic Hematopoietic Stem Cell Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: drug company is no longer making the drug
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, John Horan, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00039680; BMT Alefacept (Other: Other)
Record Dates: First submitted 2010-09-15; First posted 2011-03-22 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Thalassemia; Sickle Cell Disease; Glanzmann Thrombasthenia; Wiskott-Aldrich Syndrome; Chronic-granulomatous Disease; Severe Congenital Neutropenia; Leukocyte Adhesion Deficiency; Schwachman-Diamond Syndrome; Diamond-Blackfan Anemia; Fanconi Anemia; Dyskeratosis-congenita; Chediak-Higashi Syndrome; Severe Aplastic Anemia
Keywords: bone marrow transplant; sickle cell disease; thalassemia; Glanzmann thrombasthenia; Wiskott-Aldrich syndrome; chronic-granulomatous disease; severe congenital neutropenia; leukocyte adhesion deficiency; Schwachman-Diamond syndrome; Diamond-Blackfan anemia; Fanconi anemia; dyskeratosis-congenita; Chediak-Higashi syndrome; severe aplastic anemia
MeSH Terms: conditions — Thalassemia; Anemia, Sickle Cell; Thrombasthenia; Wiskott-Aldrich Syndrome; Granulomatous Disease, Chronic; Neutropenia, Severe Congenital, Autosomal Recessive 3; Leukocyte adhesion deficiency type 1; Shwachman-Diamond Syndrome; Anemia, Diamond-Blackfan; Fanconi Anemia; Dyskeratosis Congenita; Chediak-Higashi Syndrome; Anemia, Aplastic | interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alefacept (Experimental): Pediatric subjects with non-malignant diseases (NMD) will receive pre-conditioning with alefacept 0.5 mg/kg/dose i.v. with the first dose split on days -40 and -39 and the remaining doses given on days -33, -26, -19, and -12 (e.g. weekly for 5 doses).
  Interventions: Drug: Alefacept

INTERVENTIONS:
Drug: Alefacept — 0.25 mg/kg IV on day -40 and day -39 0.5 mg/kg IV on days -33, -26, -19 and -12 Alefacept was diluted in sterile water (2 ml total volume) and administered via i.v. push followed by a normal saline flush per package insert.
  Other Names: Amevive

SUMMARY:
Allogeneic blood and marrow transplantation remains the only viable cure for children who suffer from many serious non-malignant hematological diseases. Transplantation, however, carries a high risk of fatal complications. Much of the risk stems from the use of high dose radiation and chemotherapy for conditioning, the treatment administered just prior to transplant that eliminates the patients' marrow and immune system, effectively preventing rejection of the donors' cells. Attempts to make blood and marrow transplantation safer for children with non-malignant diseases by using lower doses of radiation and chemotherapy have largely failed because of a high rate of graft rejection.

In many such cases, it is likely that the graft is rejected because the recipient is sensitized to proteins on donor cells, including bone marrow cells, by blood transfusions. The formation of memory immune cells is a hallmark of sensitization, and these memory cells are relatively insensitive to chemotherapy and radiation. Alefacept, a drug used to treat psoriasis, on the other hand, selectively depletes these cells. The investigators are conducting a pilot study to begin to determine whether incorporating alefacept into a low dose conditioning regimen can effectively mitigate sensitization and, thereby, prevent rejection of allogeneic blood and marrow transplants for multiply transfused children with non-malignant hematological diseases.

DETAILED DESCRIPTION:
There are a large number of serious non-malignant diseases of childhood, most of them congenital and rare, which can be corrected by HSCT. These diseases are all characterized by deficiencies, either in number or in function, of marrow derived cells. These diseases usually affect immune or blood cells and frequently involve transfusion therapy with erythrocytes, platelets or granulocytes. Examples of such diseases include sickle cell disease, thalassemia major, Glanzmann thrombasthenia, Wiskott-Aldrich syndrome, chronic-granulomatous disease, severe congenital neutropenia, leukocyte adhesion deficiency, Shwachman-Diamond syndrome, Diamond-Blackfan anemia, Fanconi anemia, dyskeratosis-congenita, Chediak-Higashi syndrome, and severe aplastic anemia.

Allogeneic blood HSCT, whether performed for a malignant or a non-malignant condition, relies on the use of a pre-transplant conditioning regimen. Traditionally, very high doses of chemotherapy or total body irradiation have been utilized as conditioning. The use of intensive conditioning, which, practically speaking eliminates the host marrow and immune system, however, can produce serious and sometimes fatal infections and injuries to vital organs, such as the liver and lung. In children, the use of intensive conditioning can also produce serious late effects, including hypogonadism, stunted growth, impaired cognitive development and secondary malignancies.

Over the past decade, there has been a move to minimize the risk for such complications by reducing the intensity of conditioning regimens. Added impetus for reducing conditioning intensity arose from the observation in transplantation for thalassemia and sickle cell disease that sustained mixed chimerism, that is partial donor engraftment, is usually sufficient to cure non-malignant diseases. This observation suggested that sustained engraftment could be achieved without "ablation" or elimination of the host marrow. Pre-clinical studies demonstrated in small and large animals that sustained mixed chimerism can be achieved with preparative regimens consisting of TBI doses as low as 100-300 cGy (by comparison, standard intensity regimens typically employ 1000 cGy or more in combination with chemotherapy).

This approach was first translated in a clinical trial involving 45 adults with hematological malignancies who were not candidates for standard conditioning because of older age or serious co-morbidities. Using a single 200 cGy dose of TBI, sustained engraftment was achieved in 80% of cases and, remarkably, transplant related mortality was only 6.7% in this frail group of patients at 14 months. It is also notable that these transplants were performed primarily in the outpatient setting-the median length of hospitalization was 1 day. Low-dose TBI based conditioning has also been safely and effectively utilized for infants and children with severe combine immune deficiency and other severe immune deficiencies, undergoing related and unrelated donor transplantation. This clinical experience strongly suggests that if an effective low-dose TBI conditioning regimen can be developed for children with non-malignant diseases it could transform BMT from a costly, highly morbid, and sometimes life-taking procedure to a relatively inexpensive, safe and well-tolerated one.

Thousands and thousands of children around the world suffer from sickle cell disease and thalassemia major. There is a myriad of other less common serious non-malignant hematological diseases, which have even more devastating effects, for which HSCT remains the only viable cure. Low-dose TBI based conditioning represents a minimally toxic approach to transplantation for these children-a way to overcome alloimmunization, however, is needed to make this approach more effective. Alefacept, the only currently FDA approved agent that specifically targets memory T cells, the investigators believe, holds the key to making low-dose TBI based conditioning more effective and could, thereby, dramatically alter the field of transplantation for non-malignant diseases. sustained donor engraftment needs to be developed.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between the ages of 0-21 years at the time of admission for transplant
2. Must have been transfused with at least five platelet, erythrocyte or granulocyte units (partial or full)
3. Must have one of the following diseases:

   (a) hemoglobin SS or hemoglobin SB Sβ0 thalassemia and meet one of the criteria below for having severe sickle cell disease (i) Previous central nervous system event lasting longer than 24 hours, plus objective imaging evidence of CNS vasculopathy, with or without residual neurologic findings (ii) Frequent (≥ 3 per year for 2 years) painful vaso-occlusive episodes (defined as episode lasting ≥ 4 hours and requiring hospitalization or outpatient treatment with parenteral opioids/opiates). Must have also (iii) Recurrent (≥ 3 in lifetime) acute chest syndrome events which have necessitated exchange transfusion or chronic transfusion therapy. (iv) Any combination of ≥ 3 acute chest syndrome episodes and vasoocclusive pain episodes (defined as above) yearly for 3 years. (v) Stage I or II sickle lung disease (see appendix 1) (vi) Pulmonary hypertension, measured by tricuspid regurgitant jet velocity (TRV) of greater than 2.5m/s (vii) Osteonecrosis involving multiple joints. (viii) Sickle Cell nephropathy with moderately severe renal insufficiency estimated GFR ≥30 ml/min, but ≤60 ml/min/1.73 m2 (Requires evaluation by a nephrologist). (b) Thalassemia major (c) Glanzmann thrombasthenia (d) Wiskott-Aldrich syndrome (e) Chronic-granulomatous disease (f) Severe congenital neutropenia (g) Leukocyte adhesion deficiency (h) Shwachman-Diamond syndrome (i) Diamond-Blackfan anemia (j) Fanconi anemia (k) Dyskeratosis-congenita (l) Chediak-Higashi syndrome (m) Acquired (immune; non-inherited, non-congenital) severe aplastic anemia (only patients whose best graft source is a mismatched related donor, unrelated marrow donor or cord blood unit) (n) Other inherited or congenital marrow failure syndromes complicated by severe aplastic anemia (o) Other inherited or congenital red blood cell disorders requiring monthly chronic transfusion therapy. (p) Other inherited or congenital platelet disorders resulting in at least three inpatient hospitalizations in the past two years for bleeding. (q) Other inherited or congenital granulocyte disorders resulting in at least three inpatient hospitalizations in the past two years for infection.
4. Must have an available HLA identical sibling (HLA matched related), a non-HLA identical parent or sibling who is matched at least seven of eight loci (mismatch can be at an allele or antigen level), an unrelated adult donor who is matched at least seven of eight loci (mismatch can be at an allele or antigen level) or an unrelated cord blood unit that is matched at five of six loci (A (antigen level), B (antigen level), DRB1 (allele level)) and provides a minimum pre-cryopreservation TNC dose of 5.0 x 107 TNC/kg recipient weight.

Exclusion Criteria:

1. Hemophagocytic lymphohistiocytosis or other disorder characterized by NK cell dysfunction, since alefacept's effect is mediated by NK cells.
2. Biopsy proven cirrhosis (score IV).
3. SCD chronic lung disease ≥ stage III (see appendix 1)
4. Severe renal dysfunction defined as estimated GFR of <30 ml/min.
5. Severe cardiac dysfunction defined as shortening fraction < 25%.
6. Severe neurologic impairment other than hemiplegia alone, defined as full scale IQ ≤ 70, quadriplegia or paraplegia, inability to ambulate, inability to communicate without assistive device, or any impairment resulting in decline of Lansky performance score to <50%.
7. Karnofsky or Lansky functional performance score < 50%
8. Confirmed HIV seropositivity.
9. Patient with unspecified chronic toxicity serious enough to detrimentally affect the patient's capacity to tolerate bone marrow transplantation.
10. Patient or patient's guardian(s) unable to understand the nature and risks inherent in the BMT process.
11. History of lack of compliance with medical care that would jeopardize transplant course.
12. Patient is pregnant or lactating
13. Donor who for psychological, physiologic, or medical reasons is unable to tolerate a bone marrow harvest or receive general anesthesia.
14. Donor is HIV infected.
15. Donor is pregnant
16. Hemoglobin SS, or hemoglobin Sβ0 thalassemia patient who is eligible for one of the two trials of myeloablative conditioning currently being conducted by the Aflac Center (SALT: Alternate-Donor Bone Marrow and Cord Blood Transplantation for Children with High-Risk Sickle Cell Disease Busulfan, fludarabine, ATG and Reduced-Dose Cyclophosphamide Conditioning for Allogeneic Hematopoietic Stem Cell Transplantation in Patients with Severe Sickle Cell Disease: a pilot study
17. Patients with thalassemia major who are eligible for any multicenter study we are participating in.
18. Patients whose best graft source is a related or unrelated donor/cord blood unit that is mismatched and the patient's HLA antibody testing (see below) demonstrates an antibody directed against the disparate HLA molecule.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Horan, MD, Principal Investigator — Emory University/Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Stenger EO, Chiang KY, Haight A, Qayed M, Kean L, Horan J. Use of Alefacept for Preconditioning in Multiply Transfused Pediatric Patients with Nonmalignant Diseases. Biol Blood Marrow Transplant. 2015 Oct;21(10):1845-52. doi: 10.1016/j.bbmt.2015.06.005. Epub 2015 Jun 19. PMID 26095669

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at the Aflac Cancer and Blood Disorders Center within Children's Healthcare of Atlanta (CHOA) from November 2010 to November 2011.
Pre-assignment Details: One subject with Fanconi Anemia (FA) received fludarabine (Flu) 25 mg/m2 on days -10 to -5 and cyclophosphamide (Cy) 10 mg/kg on days -5 to -2. The other two subjects received Flu 25 mg/m2 on days -6 to -1, Cy 50 mg/kg on day -2, and low-dose total body irradiation(TBI; 200 cGy) on day -1.
Groups:
- Alefacept: Pediatric subjects with non-malignant diseases (NMD) received pre-conditioning with alefacept 0.5 mg/kg/dose i.v. with the first dose split on days -40 and -39 and the remaining doses given on days -33, -26, -19, and -12 (e.g. weekly for 5 doses).
Period: Overall Study
Arm/Group | Alefacept
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alefacept
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7 (3.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Alefacept Pre-conditioning, Measured by Number of Subjects With Full Donor Engraftment
Description: All subjects received alefacept prior to hematopoietic stem cell transplantation and were followed up to at least two years after transplantation to ensure successful engraftment.
Time Frame: Two years post-transplant
Measure: Number; unit: participants
Arm/Group | Alefacept
Number analyzed (Participants) | 3
participants | 3

2. Secondary Outcome: Number of Participants That Expressed Grade 2 or 3 Regimen-Related Toxicity
Description: Regimen-related toxicity was measured using the Bearman criteria. The Bearman criteria grades toxicity levels at Grade 1, Grade 2, Grade 3, and Grade 4. In this system, grade I toxicity is reversible without treatment and grade 2 is not life threatening, but requires treatment. Grade 3 requires life-support intervention and grade 4 is fatal. All regimen-related toxicities were determined to be unlikely attributable to the study drug.
Time Frame: Day 42 post-transplant
Measure: Number; unit: participants
Arm/Group | Alefacept
Number analyzed (Participants) | 3
participants | 2

3. Secondary Outcome: Number of Participants That Expressed Successful Neutrophil Engraftment
Description: Neutrophil engraftment was assessed with absolute neutrophils >500*10^8/kg by 100 days post transplant. Neutrophils were counted by performing a complete blood cell count (CBC).
Time Frame: Day 100 post-transplant
Measure: Number; unit: participants
Arm/Group | Alefacept
Number analyzed (Participants) | 3
participants | 3

4. Secondary Outcome: Incidence of Greater Than or Equal to 85% CD3 Donor Chimerism
Description: CD3 chimerism was measured from peripheral blood lymphocytes 30 days post transplant. DNA chimerism analysis was performed by amplified fragment length polymorphism.
Time Frame: Day 30 post-transplant
Measure: Number; unit: participants
Arm/Group | Alefacept
Number analyzed (Participants) | 3
participants | 3

5. Secondary Outcome: Incidence of 100% CD33 Donor Chimerism
Description: CD33 chimerism was measured from peripheral blood lymphocytes 30 days post transplant. DNA chimerism analysis was performed by amplified fragment length polymorphism.
Time Frame: Day 30 post-transplant
Measure: Number; unit: participants
Arm/Group | Alefacept
Number analyzed (Participants) | 3
participants | 3

6. Secondary Outcome: Number of Participants Who Experienced Acute Graft-versus-host Disease (aGVHD), Measured by NIH Consensus Criteria (NCC) Score: Grade II-IV
Description: Cumulative Incidence of Grade II-IV aGVHD Score at 30 Days. The NIH Consensus grading and severity criteria includes physical assessments of skin, oral cavity, eyes, gynecological and laboratory data and patient reports. Each domain is scored from Grade 0 (no involvement) to Grade IV (severe involvement).
Time Frame: Day 30 post-transplant
Measure: Number; unit: participants
Arm/Group | Alefacept
Number analyzed (Participants) | 3
participants
  Grade II | 2
  Grade III | 1
  Grade IV | 0

7. Secondary Outcome: Number of Participants Who Experienced Chronic Graft-versus-host Disease (cGVHD), Measured by the NIH Criteria Consensus (NCC)
Description: The severity criteria of chronic graft-versus-host disease (cGVHD) recommended by the NIH Criteria Consensus (NCC) was employed. The number of organs involved and the severity of the disease in these organs dictated the global summary score used to define the disease as mild, moderate, or severe. Mild disease indicates one or two organs involved each with a maximal score of 1. Moderate disease indicates three or more organs involved with a score of 2 in any individual organ, or lung involvement with a score of 1. Severe global GVHD is defined by a score of 3 in any organ, or a lung score of 2.
Time Frame: Day 100 post-transplant
Measure: Number; unit: participants
Arm/Group | Alefacept
Number analyzed (Participants) | 3
participants
  Mild cGVHD | 0
  Moderate cGVHD | 1
  Severe cGVHD | 1

ADVERSE EVENTS:
Arm/Group | Alefacept
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alefacept (N=3)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Chronic graft versus host disease (Immune system disorders) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alefacept (N=3)
Pulmonary aspergillosis (Infections and infestations) | 1 (1)
Cytomegalovirus (CMV) Viremia (Infections and infestations) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bacteremia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Production of alefacept was halted in 2011.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes